CLINICAL TRIAL: NCT05860244
Title: Effect of Salbutamol on Walking Capacity in Ambulatory ALS Patients
Acronym: WALKALS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP190724
Record Dates: First submitted 2023-04-24; First posted 2023-05-16 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Walking Capacity; Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Walking capacity; Salbutamol; Ventolin
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salbutamol (Experimental): Salbutamol 2mg/5ml syrup : 2mg TID salbutamol for 3 months, then 4 mg TID for 3 months
  For each investigated dose (6 mg then 12 mg), the treatment will be titrated during a 4 days period:
  At beginning of the first 3-month period : Month 0 D1: 2mg in the morning; D2-D3: 2 mg in the morning and 2mg in the evening for two days; From D4 and until the end of first 3-month period (until the M3 follow-up visit): 2mg in the morning, at noon and in the evening
  At beginning of the second 3-month period : Month 3 D1: 4mg in the morning, 2mg at noon, 2 mg in the evening; D2: 4 mg in the morning, 2 mg at noon and 4mg in the evening; J4 and for 3 months (until the M6 follow-up visit) : 4mg in the morning, at noon and in the evening.
  Interventions: Drug: Salbutamol
- placebo of salbutamol (Placebo Comparator): Placebo syrup : 2mg TID salbutamol for 3 months, then 4 mg TID for 3 months
  For each investigated dose (6 mg then 12 mg), the treatment will be titrated during a 4 days period:
  At beginning of the first 3-month period : Month 0 D1: 2mg in the morning; D2-D3: 2 mg in the morning and 2mg in the evening for two days; From D4 and until the end of first 3-month period (until the M3 follow-up visit): 2mg in the morning, at noon and in the evening
  At beginning of the second 3-month period : Month 3 D1: 4mg in the morning, 2mg at noon, 2 mg in the evening; D2: 4 mg in the morning, 2 mg at noon and 4mg in the evening; J4 and for 3 months (until the M6 follow-up visit) : 4mg in the morning, at noon and in the evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol — Salbutamol for 6 months
  Arms: Salbutamol
Drug: Placebo — Placebo Syrup for 6 months
  Arms: placebo of salbutamol

SUMMARY:
Preclinical and clinical data strongly suggest that administration of salbutamol in ALS patients may improve walking capacity related to motor fatigue by enhancing neuromuscular transmission. Salbutamol may exert a neuroprotective effect and slow down the progression of clinical signs and symptoms. The main objective of the study is to test the efficacy of salbutamol on walking capacity in ALS patients and the secondary objective is to measure the target engagement of salbutamol on the neuromuscular junction (NMJ) at EMG (decrement of repetitive nerve stimulation in three nerves/muscle couples), as well as safety and tolerability. The exploratory objectives are to study the effect of salbutamol on fatigue scales, muscle strength, respiratory function, motor unit count, muscle and spinal MRI parameters and blood biomarkers

DETAILED DESCRIPTION:
Based on a strong preclinical and clinical rationale the main hypothesis is that the administration of salbutamol in ALS patients may improve the walking capacity related to motor fatigue by enhancing the neuromuscular transmission. Salbutamol may also exert a neuroprotective effect and slow down the progression of clinical signs and symptoms.

To test these hypotheses, the investigator team will implement a monocentric, randomized, controlled, pilot study to evaluate the effect of salbutamol on walking capacity in ambulatory ALS patients with a total duration of 24 months and a treatment period of 6 months for each patient. The project Team will use as secondary and exploratory endpoints target engagement and efficacy up-to date biomarkers such as quantitative muscle strength evaluation, functional neuromuscular evaluation and spinal and muscle MRI. Tolerability and safety will also be studied. Salbutamol has been used for a long time and is usually well tolerated. The objective of the study is to evidence a signal of efficacy paving the way for a confirmatory phase 3 trial.

In parallel to this, the use of muscle and spinal MRI as well as of quantitative muscle strength evaluation as exploratory endpoints will pave the way to their development as biomarkers of disease progression in ALS. Thanks to the data collected in this study, the team will give proof of their accuracy, with a view to ameliorate the prognostication and monitoring of disease progression and survival, as well as to improve the understanding of the interaction between muscular and central degeneration. A further aim of this study will be to provide a proof of concept that spinal and muscle MRI can constitute a biomarker of the efficacy of investigational drugs targeting muscles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the revised El Escorial criteria for probable or definite sporadic ALS
* Adult patients between 18 and 75 years of age
* Patients who are ambulatory and able to perform the 6MWT and quantitative muscle testing at screening (ALSFRS-R-walking = 3)
* Patients able and willing to travel to the site, and, in the investigator's opinion, who are likely to attend visits for at least 6 months
* Patients who signed written informed consent
* Stable dose of riluzole for a minimum of 4 weeks prior to baseline or has not taken it for 4 weeks prior to baseline
* For child-bearing aged women, efficient contraception (cf protocol p32)
* Forced vital capacity (fVC) in a sitting position > 70 %

Exclusion Criteria:

* Patients with significant spasticity of the lower limbs interfering with walking capacity (Ashworth scale score > 2)
* Patients with fronto-temporal dementia associated with ALS
* Patients presenting respiratory insufficiency causing dyspnea during walking
* Patients taking drugs that could interfere with NMJ function (anticholinesterase …) or muscle function (steroids, statins…)
* Patients taking any forbidden drugs (see list in annex)
* Hypersensitivity to salbutamol or to excipients of the drug and placebo
* Known contraindication for the studied drug such as ischemic cardiomyopathy or risk of ischemic cardiomyopathy: history of ischemic heart disease or coronaropathy or/and significant ischemic ECG alterations at screening visit
* Any clinically significant alterations in the following biological parameters glycemia, kalemia, creatinemia and hematology in the month prior to inclusion according to local laboratory threshold (cf protocol page 33)
* Vulnerable persons defined in Articles L1121-5 to L 1121-8-1 and L1122-1-2 of the Code de la Santé Publique* (*CSP)
* Participation in another interventional trial up to 3 months before inclusion
* Patients having any relevant concomitant disease considered at risk of interfering with study procedures in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
walking capacity | Month 6
  6 minutes walking test distance (6MWT)
walking capacity | Month 3
  6 minutes walking test distance (6MWT)

SECONDARY OUTCOMES:
Target engagement: | baseline, month 3, month 6
  percentage of change of the decrement at electromyography after repetitive nerve stimulation.
functional quantitative decline description over time in ALS patients | baseline, month 3, month 6
  Revised ALS Functional Rating Scale-r (ALSFRS-r) composed by 12 questions scoring from 0 to 4 with a maximal score of 48
walking scale | baseline, month 3, month 6
  Twelve items Multiple Sclerosis (MS) Walking Scale (12-MSWS) ( score: 5 to 60 ( severe difficulty)) . Walking improvement on the MSWS-12 is indicated by negative change scores.
Fatigue and depression scale | baseline, month 3, month 6
  Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. ( score : 9 (no fatigue ) to 63 (extreme fatigue)
Respiratory assessment | baseline, month 3, month 6
  Forced Vital Capacity (FVC): the maximum amount of air that a person can exhale as hard and as long as possible from the lungs after a maximum inspiration and Forced Expiratory Volume in the first second of exhalation (FEV1) : FEV1 is the most frequently used index for assessing airway obstruction, bronchoconstriction or bronchodilation
Thigh muscle volume | baseline, month 3, month 6
  bioelectrical impedance analysis (BIA)
Muscle volume | baseline, month 3, month 6
  Muscle MRI in cm3
Biomarkers of muscle damage | baseline, month 3, month 6
  CPK, LDH and creatinine serum levels
Quality of life scale | baseline, month 6
  The Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) ( score: 0 to 160 bad quality of life)
Motor unit number | baseline, month 6
  Motor unit count (MUNIX method)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No